CLINICAL TRIAL: NCT05923203
Title: Binaural Cue Sensitivity in Children and Adults With Combined Electric and Acoustic Stimulation
Brief Title: Combined Electric and Acoustic Hearing (EAS) in Children and Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hearts for Hearing (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, René Gifford, Chief of Audiology and Research, Hearts for Hearing
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 222052; 1R01DC020194-01A1 (NIH)
Record Dates: First submitted 2023-06-07; First posted 2023-06-28 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-04

CONDITIONS: Cochlear Implant; Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Electricity; Acoustic Stimulation; Technology; Hearing Aids

STUDY DESIGN:
Intervention Model Description: There will be four groups of study participants including two experimental groups (pediatric and adult EAS) as well as two control groups [pediatric and adult listeners with normal hearing (NH).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adult use of EAS (Experimental): Clinical intervention; Adults with CI and the fitting of electric and acoustic stimulation (EAS) technology in the implanted ear(s).
  Interventions: Other: Electric and acoustic stimulation (EAS) technology in the implanted ear(s)-this is the combination of a cochlear implant (CI) and hearing aid (HA) in the implanted ear(s)
- Pediatric use of EAS (Experimental): Clinical intervention; Children with CI and the fitting of electric and acoustic stimulation (EAS) technology in the implanted ear(s).
  Interventions: Other: Electric and acoustic stimulation (EAS) technology in the implanted ear(s)-this is the combination of a cochlear implant (CI) and hearing aid (HA) in the implanted ear(s)
- Children with Normal Hearing (No Intervention): Children with normal hearing; acoustic only
- Adults with Normal Hearing (No Intervention): Adult with normal hearing; acoustic only

INTERVENTIONS:
Other: Electric and acoustic stimulation (EAS) technology in the implanted ear(s)-this is the combination of a cochlear implant (CI) and hearing aid (HA) in the implanted ear(s) — This is a clinical fitting of an FDA approved EAS system for study participants that have received or who are scheduled to receive a CI based on clinical recommendations (i.e. not study related). The investigators will activate the CI sound processor's integrated HA circuit to allow for low-frequency acoustic amplification and mid-to-high frequency electric stimulation in the implanted ear(s) using recommended and accepted clinical practices and audiologic verification. EAS fitting will be completed using FDA approved clinical software and thereby is within the electrical and clinical specifications of the FDA approved device and accompanying software.
  Arms: Adult use of EAS; Pediatric use of EAS

SUMMARY:
Cochlear implants are surgically implanted devices which restore the ability to hear to the hearing impaired. Improvements in surgery and electrodes have results in an increased number of adults and children who have residual hearing and can benefit from electric and acoustic hearing in the same ear. This is called Electric Acoustic Stimulation (EAS). Many studies have shown that adult EAS users show significant benefits for speech understanding in noise and spatial hearing tasks as compared to a CI paired only with a contralateral HA. Even though this type of hearing is becoming more common, there is limited research on how it can be beneficial to children with CIs. The benefits of this study are a greater understanding of the participant's speech understanding, binaural processing, and spatial hearing. The results will help audiologists and researcher better understand how cochlear implants work, specifically when using electric and acoustic hearing in the same ear.

DETAILED DESCRIPTION:
Cochlear implantation with minimally traumatic surgical techniques and atraumatic electrode arrays has led to an increasing prevalence of adult and pediatric cochlear implant (CI) recipients with the potential for combined Electric and binaural Acoustic Stimulation (EAS). Many studies have demonstrated that adult EAS users consistently exhibit significant benefits for speech understanding in noise and spatial hearing tasks as compared to a CI paired only with a contralateral HA. Research has also demonstrated that sensitivity to interaural time difference (ITD) and interaural level difference (ILD) cues is correlated with EAS benefit for postlingually deafened adult listeners. Despite this active phase of discovery, there is still a striking paucity of research on EAS outcomes in pediatric CI users, the expected trajectory of benefit following EAS fitting, as well as underlying mechanisms driving EAS benefit (or lack thereof) in all populations. There is a disconnect between EAS availability and EAS utilization in all CI recipients and current audiological management of EAS candidates is not data driven. This is problematic given the protracted maturation of the binaural system and the fact that researchers do not understand what additional effects sensorineural hearing loss and combined EAS may have on the developing binaural system. The proposed research activities will describe the time course of binaural development using behavioral and objective responses to interaural differences in timing (phase) and level as well as allow for a natural factor investigation of a clinical intervention, the EAS fitting, on said development. Within the context of a clinical trial, the investigators will compare acute and chronic EAS outcomes for speech recognition and spatial hearing as related to binaural cue sensitivity, cue weightings and underlying neural synchrony necessary for ITD resolution. The investigators have proposed a single-group assignment for both adult and pediatric EAS users and will also include chronological- and hearing-age-matched listeners with normal hearing (NH). A within-subjects, accelerated longitudinal design for both EAS and NH listeners will provide insight into the developmental trajectory of the binaural system for children NH and will provide a benchmark for interpreting effects of sensorineural hearing loss, asymmetry in audibility resulting from cochlear implantation, and EAS use on said trajectory. Our proposed research activities will help close the gap between what is technologically possible with EAS technology and what is clinically implemented by otologists and audiologists investigating development of binaural sensitivity and spatial hearing abilities. The resultant data will comprise the first comprehensive description of behavioral and electrophysiologic measures of binaural hearing in adults and children both with NH and EAS and will uncover information about our EAS clinical populations holding high potential for clinical application in device fittings as well as audiologic and otologic clinical recommendations regarding cochlear implantation.

AIM 1: Emergence of binaural cue sensitivity in EAS users. The investigators will investigate emergence of binaural sensitivity for ITD and ILD cues as well as ITD/ILD cue weighting, which is critical for children with developing binaural function and underlying neural synchronization. Hypotheses: 1a) Pediatric EAS users will demonstrate an emergence of binaural cue sensitivity following a period of chronic EAS use incorporating bilateral LF acoustic amplification, 1b) there will be a relationship between listener age and ITD/ILD weighting for lateralization with the youngest EAS candidates assigning greater weight to ILDs due to immaturities in neural synchronization, and 1c) the time course of pediatric acoustic ITD/ILD development will be correlated with absolute and interaural auditory sensitivity for LF acoustic hearing.

AIM 2: Degree and time course of EAS benefit for speech and spatial discrimination informed by behavioral and objective estimates of binaural cue utilization. The investigators will describe EAS listener performance (CI+HAbilat) and EAS benefit (CI+HAbilat - CI+HAcontra) for (1) tasks of speech recognition in co-located, diffuse, and spatially separated noise, and (2) tasks of spatial discrimination. The investigators will relate these to ITD/ILD sensitivity measured both behaviorally (Aim 1) and electrophysiologically (Aim 2) via cortical auditory evoked potentials (CAEPs) reflecting brainstem-initiated processes inherited by the central auditory system. Hypotheses: 2a) EAS benefit will be observed for speech recognition and spatial discrimination with chronic EAS use, which will be mediated by access to LF ITD cues estimated via both behavioral and objective measures, and 2b) there will be a relationship between behavioral and objective measures of binaural cue utilization and EAS benefit for speech recognition and spatial hearing.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 5 to 17 years of age with either normal hearing (n=40) or at least 1 cochlear implant (CI) and binaural low-frequency acoustic hearing (n=40); adults aged 18+ years with either normal hearing (n=40) or at least 1 CI and binaural low-frequency acoustic hearing (n=40).
2. Experimental participants must have at least one CI and bilateral mild to severe sensorineural hearing loss For CI participants, audiometric thresholds in the non-CI ear must be consistent with at least a mild sensorineural hearing loss; that is, the investigators will not be enrolling participants with single-sided deafness (SSD) For CI participants, unaided audiometric thresholds must be less than or equal to 80 dB HL for 125 and 250 Hz, in both ears.
3. Nonverbal cognitive abilities within the typical range for all participants; adult participants must also pass cognitive screening via Montreal Cognitive Assessment (MoCA or HI-MoCA).
4. No confounding diagnosis such as autism, auditory neuropathy, neurological disorder, or general cognitive impairment.
5. Willingness to use EAS technology in the implanted ear(s) to be verified via data logging from cochlear implant and hearing aid software.

Exclusion Criteria:

1. Nonverbal intelligence standard score < 85 (for any participant).
2. MoCA or HI-MoCA score < 26 for adult participants.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in BEL sentence score demonstrating EAS benefit for speech recognition in noise (CIHA+HA - CI+HA) | This will be measured at multiple time points including at or within 1 month of EAS activation (adults & peds), 6 months (adults & peds), 12 months (adults & peds, and 24 months (peds)
  Speech recognition will be assessed with co-located (S0N0) and spatially separated noise (S0N90 and S0N270) using the BEL sentences with two different male or female talkers as the maskers. Target speech will be fixed at 70 dB SPL for both speech stimuli and the investigators will assess performance for two listening conditions: CI+HA and CIHA+HA.
Change in BKB-SIN score demonstrating EAS benefit for speech recognition in noise (CIHA+HA - CI+HA) | This will be measured at multiple time points including at or within 1 month of EAS activation (adults & peds), 6 months (adults & peds), 12 months (adults & peds, and 24 months (peds)
  Speech recognition will be assessed with co-located (S0N0) and spatially separated noise (S0N90 and S0N270) using the BKB-SIN test with multi-talker babble as the masker. Target speech will be fixed at 70 dB SPL for both speech stimuli and the investigators will assess performance for two listening conditions: CI+HA and CIHA+HA.

SECONDARY OUTCOMES:
EAS benefit for minimal audible angle (MAA) (CIHA+HA - CI+HA) | This will be measured at multiple time points including at or within 1 month of EAS activation (adults & peds), 6 months (adults & peds), 12 months (adults & peds, and 24 months (peds)
  MAA thresholds will be obtained by presenting 2 successive stimuli from different positions in the horizontal plane and requesting that the listener indicate whether the 2nd stimulus was to the left or to the right of the standard. Noise stimuli will include a BBN (100-8000 Hz) and LF noise (100-800 Hz). Three listening conditions will be tested: 1) bilateral HA (HA+HA), 2) bimodal (CI+HA), and EAS (CIHA+HA).
ITD sensitivity | This will be measured at multiple time points including at or within 1 month of EAS activation (adults & peds), 6 months (adults & peds), 12 months (adults & peds, and 24 months (peds)
  ITD thresholds will be measured using tonal and noise-band carriers. This task will be completed using both acoustic and electric stimulation with the latter achieved via direct connection to the CI sound processor allowing for investigation of binaural interference.
ILD sensitivity | This will be measured at multiple time points including at or within 1 month of EAS activation (adults & peds), 6 months (adults & peds), 12 months (adults & peds, and 24 months (peds)
  ILD thresholds will be measured using tonal and noise-band carriers. This task will be completed using both acoustic and electric stimulation with the latter achieved via direct connection to the CI sound processor allowing for investigation of binaural interference.

CONTACTS AND LOCATIONS:
Overall Officials: René H Gifford, PhD, Principal Investigator — Hearts for Hearing
Locations (4):
- United States (4):
  - Hearts for Hearing, Edmond, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University Of Texas at Austin, Austin, Texas
  - University Of Wisconsin Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT05923203/Prot_SAP_001.pdf